CLINICAL TRIAL: NCT07079020
Title: Multicenter Cohort Study on Efgartigimod for Consolidation Therapy After the Acute Exacerbation of Generalized Myasthenia Gravis in Adults
Brief Title: Efgartigimod for Consolidation Therapy in gMG
Status: Not yet recruiting | Type: Observational
Sponsor: Da, Yuwei, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: LYS[2025]190-002
Record Dates: First submitted 2025-06-29; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Efgartigimod+SOC: Initiate efgartigimod combined with standard of care (SOC) therapy according to the protocol within one month after consolidation baseline.
- SOC: No additional treatments are to be administered other than the standard of care (SOC) therapy.

SUMMARY:
The goal of this observational study is to evaluate the efficacy and safety of consolidation therapy with corticosteroids and/or immunosuppressants combined with efgartigimod in patients with generalized myasthenia gravis after the acute exacerbation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female.
2. Diagnosis of myasthenia gravis (MG) based on the following:

   1. Typical clinical features of MG.
   2. At least one of the following:

   Seropositive for anti-AChR antibodies (confirmed by reliable assay). Abnormal neuromuscular transmission on electrophysiological testing (e.g., RNS or SFEMG).

   Positive neostigmine test or documented response to cholinesterase inhibitors.
3. MGFA classification II-IV at consolidation baseline.
4. Seropositive for anti-AChR antibodies (required for enrollment).
5. Hospitalized for myasthenic crisis (MC) in the acute exacerbation and completed one treatment cycle of efgartigimod: acute exacerbation definition: Presence of MC warning signs (new or worsening within 2 weeks): Bulbar symptoms: Dysphagia, choking, weak cough, dysarthria. Respiratory symptoms: Dyspnea, respiratory muscle weakness. Generalized weakness: Head drop, jaw weakness, facial weakness. One treatment cycle of efgartigimod: 10 mg/kg IV, once weekly for 4 doses.
6. ≥2-point improvement in MG-ADL score from acute exacerbation baseline by Day 4 of efgartigimod treatment.
7. Willing and able to provide written informed consent before study participation.

Exclusion Criteria:

1. Treatment with IVIg, plasma exchange (PE), IV methylprednisolone (IVMP), or immunoadsorption (IA) within 1 month before consolidation baseline.
2. Thymectomy within 6 months before exacerbation baseline.
3. Use of immunomodulatory monoclonal antibodies or investigational drugs (not listed above) within 3 months before baseline or 5 half-lives (whichever is longer).
4. Pregnancy or lactation (women of childbearing potential must have negative pregnancy test and use contraception).
5. Known hypersensitivity to efgartigimod or any FcRn-targeting therapy.
6. Clinically significant comorbidities, including severe cardiovascular, hepatic, renal, pulmonary, or hematologic disorders, active malignancy and uncontrolled systemic infections.
7. Other autoimmune diseases that may interfere with efficacy assessment (e.g., uncontrolled thyroid disease, severe rheumatoid arthritis).
8. Any other condition deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AChR antibody-positive adults with generalized myasthenia gravis who responded to acute exacerbation treatment and underwent consolidation therapy
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving and maintaining minimal symptom expression (MSE) for at least 4 months after first attaining MSE status at any time during the consolidation therapy period within 2 months. | Consolidation baseline up to Month 6
  The MG-ADL is an 8-item patient-reported scale to assess MG symptoms and their effects on daily activities. The scale comprises 2 items on daily life activities and 6 items on symptoms. The MG-ADL total score range is 0-24, with higher scores indicative of greater disease severity. A patient was considered achieving MSE if there was a 1 or 0 on the MG-ADL total score ≥4 consecutive months after first attaining MSE status at any time during the consolidation therapy period within 2 months.

SECONDARY OUTCOMES:
Proportion of patients achieving both minimal symptom expression (MSE) and a daily corticosteroid dose ≤5 mg at Month 12. | Consolidation baseline up to Month 12
  The MG-ADL is an 8-item patient-reported scale to assess MG symptoms and their effects on daily activities. The scale comprises 2 items on daily life activities and 6 items on symptoms. The MG-ADL total score range is 0-24, with higher scores indicative of greater disease severity. A patient was considered achieving MSE if there was a 1 or 0 on the MG-ADL total score.
Proportion of patients with MGFA Post-Intervention Status (MGFA-PIS) at Month 6 and Month 12 | Consolidation baseline up to Month 6 AND Month 12
Change from baseline in MG-ADL scores at Month 6 and Month 12 | Consolidation baseline up to Month 6 AND Month 12
  The Myasthenia Gravis Activities of Daily Living (MG-ADL) is an 8-item patient-reported scale to assess MG symptoms and their effects on daily activities. The scale comprises 2 items on daily life activities and 6 items on symptoms. The MG-ADL total score range is 0-24, with higher scores indicative of greater disease severity.
Change from baseline in QMG scores at Month 6 and Month 12 | Consolidation baseline up to Month 6 AND Month 12
  The Quantitative Myasthenia Gravis (QMG) scale quantifies disease severity based on impairments of body functions and structures as defined by the International Classification of Disability and Health. The QMG scale consists of 13 items that measure endurance or fatigability, and accounts for fluctuations in disease state. The QMG total score range is 0-39, with higher scores indicative of greater disease severity.
Proportion of patients achieving minimal symptom expression (MSE) at Month 6 | Consolidation baseline up to Month 6
Proportion of patients achieving minimal symptom expression (MSE) with daily corticosteroid dose ≤5 mg at Month 6 | Consolidation baseline up to Month 6
Incidence of acute exacerbations, impending myasthenic crisis, or myasthenic crisis events during the study period | Consolidation baseline up to Month 12
Types and frequencies of adverse events (AEs) and serious adverse events (SAEs) during the study period | Consolidation baseline up to Month 12